CLINICAL TRIAL: NCT06117059
Title: The PRECISION Study: A Phase II Study of 3 Fractions of Prostate SBRT With RayPilot System and HypoCath Image Guidance for Men With NCCN Low or Intermediate Risk Prostate Cancer
Brief Title: The PRECISION Study: 3 Fractions of Prostate SBRT and RayPilot HypoCath Image Guidance
Acronym: PRECISION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC23118
Record Dates: First submitted 2023-10-10; First posted 2023-11-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Localized Prostate Cancer; Low Risk Prostate Cancer; Intermediate Risk Prostate Cancer
Keywords: SBRT; SABR; PROSTATE CANCER; RayPilot; HypoCath; Continuous tracking; 3 fractions
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm Phase II study of 3 fractions of prostate SBRT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 fractions of prostate Stereotactic Body Radiotherapy (SBRT) (Experimental): 3 fractions of SBRT with image guidance using the RayPilot HypoCath system given on 3 consecutive days
  Interventions: Radiation: 3 fractions of prostate SBRT

INTERVENTIONS:
Radiation: 3 fractions of prostate SBRT — Radical radiotherapy using only 3 fractions of prostate SBRT over 3 consecutive days

SUMMARY:
The investigators want to investigate whether it is possible to reduce the number of curative radiotherapy doses from 5 to only 3 for men with localized early prostate cancer. The aim of the study is to ensure that the side effects of the 3-dose treatment are the same or potentially lower than those already published when using the 5-dose treatment as used in the UK PACE-B trial (NCT01584258). The name of this type of radiotherapy is Stereotactic Body Radiotherapy (SBRT) or participants may see it referred to as Stereotactic Ablative Radiotherapy (SABR). The study is a two-stage single arm Phase II study open to those Centres that use the RayPilot HypoCath tumour tracking system (Micropos Medical). This commercially available system was not available at the time of the original PACE-B study. The system acts like a Global Positioning Device (GPS) to continuously track the prostate position during radiotherapy. If the prostate moves more than 2mm (about 0.08 in) from its intended position during the treatment, then the radiotherapy team are alerted, and the treatment halted until the prostate moves back into the correct position. The ability to understand exactly where the prostate is throughout the treatment ensures the intended dose hits the cancer and does not accidentally increase the dose to the nearby bladder and rectum. The system is a modification of a standard urinary catheter which sits within the bladder with the GPS placed within the wall of the catheter as it passes through the prostate. The investigators are not testing the system as it is commercially available but using it to improve the accuracy of radiotherapy delivery, reducing the number of days of treatment, minimizing side effects and helping ease the burden on busy radiotherapy Departments.

DETAILED DESCRIPTION:
Prostate cancer is the commonest male cancer and sadly more than 10,000 men die each year from the disease in the UK. This is actually a greater number than women who die from breast cancer each year in the UK. If diagnosed at an early stage, the chances of being cured of the disease are high through either surgery (prostatectomy) to remove the prostate or through radiation treatment (radiotherapy). Both treatment options are associated with quality of life changing impacts on sexual, bowel and bladder function, with survivors having to manage these side effects for the rest of their lives. It is a key area of research to try and identify who may be at particular risk and to minimize these risks. The development of increasingly sophisticated radiotherapy machines (linear accelerators) which can deliver radiotherapy more precisely has allowed the radiotherapy for prostate cancer to be transformed over the last decade. The number of treatments required for cure has been reduced from 39 over nearly 8 weeks, to 20 over 4 weeks, and more recently to only 5 over 1-2 weeks, greatly improving patient convenience through less travel, days off work, or time in hospital away from loved ones. Importantly technology has reduced but not removed the risk of both initial and then longer term permanent side effects.

In this study the investigators want to reduce the number of treatments down to only 3, given on consecutive days, further enhancing the patient experience and providing evidence that this number of treatments could become the new standard of care. In this study the investigators will be using the very latest state of the art radiotherapy machines and the unique RayPilot system, adopted for routine use by a small number of global radiotherapy centres when delivering prostate SBRT(Stereotactic Body Radiotherapy). The ability to track the position of the prostate cancer throughout the radiotherapy treatment using RayPilot allows the treatment to be given more precisely with less dose being given to the surrounding bladder and rectum. It also ensures that all the intended dose is given to the cancer as the treatment can be interrupted should the cancer move due to rectal gas, changes in bladder filling or simply the patient moving position on the treatment bed, maximizing the chances of cure and minimizing the risk of life changing side effects.

This is a single arm 2 stage Phase II study that will test the safety of the 3 fraction radiotherapy schedule. It has built in safety measures to ensure that the immediate post treatment side effects on the bowel and bladder are within the expected limits of acceptance at 12 weeks post completion of treatment. After 43 patients are recruited the initial data will be analyzed and if acceptable the study will continue until all 100 patients have been recruited. The study will be opened in the UK with Edinburgh as the lead Centre, and also in a number of other global centres each of which will ask for their own local ethical approval and sponsorship. The anonymized data from each Centre will be recorded on a trial specific RedCap database held by the University of Edinburgh for analysis of the trial results.

On the day of treatment planning, the patient will be met by the research team and taken to the MRI suite. Patients will have already have been prescribed a rectal suppository by their GP to bring with them. The patient will be directed to the toilet at the MRI scanner and will pass the suppository into their rectum and wait 30 seconds before evacuating it. The aim is to dispel rectal gas not necessarily to move the bowels. Patients will also empty their bladder of urine. The research nurse or radiographer will then place a dummy RayPilot HypoCath (called a ViewCath) or a simple standard Foley urinary catheter if preferred, and fill the bladder with 100-150 mls of water. This volume is recorded and kept as a constant for each day of subsequent treatment. An MRI of the prostate is then performed with standard T1 and T2 anatomical images and functional Dynamic Contrast Enhanced (DCE) and diffusion weighted (DW) sequences that identify the tumour. The MRI scan will last approximately 20minutes. On completion the patient is then taken for the planning CT scan within the Radiotherapy Department. The bladder is drained and then refilled through the catheter to the same volume as the MRI scan. The suppository is only repeated if there has been a substantial change in the rectal volume between the MRI and planning CT scan. The CT scan takes 15 minutes and then the patient has the catheter removed and is free to go home.

The MRI and CT scan are fused together to allow the clinician to plan the radiotherapy treatment on the radiotherapy planning computer system. Once the target and surrounding normal tissues have been outlined and a radiotherapy plan developed then the patient is ready to start treatment. The planning of treatment takes 2 weeks on average.

On the day of treatment the patient will be met in the Radiotherapy Department by the research team and taken to the treatment machine. A baseline PSA (Prostate Specific Antigen) should have been taken prior to the start date however if not then this blood test will be performed by the research team. A baseline quality of life patient reported outcome measure (PROM) consisting of IPSS (International Prostate Symptom Score), EPIC-26 (Expanded Prostate Cancer Index Composite), EIIF-5 (International Index of Erectile Function), Vaizey Score (A measure of bowel symptoms including incontinence)and clinician assessed RTOG (Radiotherapy and Oncology Group)and CTCAE (Common Terminology Criteria for Adverse Events) bowel and bladder toxicity scores taken. These forms will take approximately 20 minutes to complete.

The patient will then use a rectal suppository in the toilet as per the planning scans and empty their bladder. The research team will then place the RayPilot HypoCath into the bladder under local anesthetic. This procedure is no different to placing a normal Foley urinary catheter. The bladder will be filled with the same volume of water used at the time of the planning scans and is then ready for treatment.

Patients lie on their back in the linear accelerator on a special RayPilot receiver couch top with their ankles resting on foot stocks to reduce movement. The patient is set up for treatment as per standard of care when delivering prostate SBRT. A check cone beam CT scan taken by the linear accelerator is taken to verify the treatment position and that the prostate is correctly within the radiotherapy field. If this is correct the treatment beam is switched on and treatment starts. Should the prostate move beyond the 2mm level of tolerance set for the treatment then the beam is interrupted and restarted when the prostate has returned to the correct position. If needed a repeat cone beam treatment CT may be taken before the beam is switched on should the prostate fail to settle back into position and the patients new treatment position used. The time taken to deliver the treatment from entering the linear accelerator to leaving the room is 20-30 minutes. On completion of the first day of treatment the patient drains the bladder and a flip flow valve placed on the end of the RayPilot HypoCath to allow the patient to continue to pass urine as needed by simply opening the valve and letting the bladder drain through the catheter into the toilet.

The patient will start their treatment on a Tuesday if possible and be treated on 3 consecutive days in total. On day 2 and 3 the treatment procedure is identical to the day 1. On completion of treatment on day 3 the HypoCath is removed and repeat RTOG and CTCAE toxicity and an IPSS assessment taken by the research team before the patient goes home.

The patients are then followed up in the outpatient clinical by the research team and the follow up PSA and toxicity assessments are made. The follow up schedule is weeks, 2, 4, 8 and 12 post treatment, and then months 6, 9, 12, 18 and 24 before they then leave the study. Prior to each visit the local GP/ Community practice will have taken the PSA blood test to assess tumour response. If this has not been done prior to clinic then it will be taken by the research team in the clinic. PSA blood tests at FU are standard procedure and the interval is the same as men treated by prostate SBRT who are not in the study except for an extra visit at weeks 2 and month 9 for this study.

The level of acute radiotherapy side effects up to and including week 12 will be assessed as follows RTOG/CTCAE & IPSS weeks 2, 4, 8, 12 EPIC-26 & Vaizey Score weeks 4 and 12 IIEF-5 week 12. The anticipated length of each clinic visit will be 20 minutes The level of late persistent radiotherapy side effects up to and including month 24 be asses as follows RTOG/CTCAE, IPSS, EPIC-26 & VAIZEY Score at months 6,9, 12, 18, 24 IIEF-5 at months 6, 12 and 24 only. After 24 months patients will leave the study and be followed up within the Departmental follow up policy for long term outcome data

ELIGIBILITY:
Inclusion Criteria:

* low and favorable intermediate NCCN Criteria patients
* Prostate volume under 80cc
* IPSS under 20
* Q-max above 10cc per second and urinary residual less than 150mls
* No TURP
* No hip replacements
* No previous radiotherapy to the pelvis
* No active second malignancy except skin SCC or BCC for the last 2 years
* No history of inflammatory bowel disease
* No co-morbid illness that would make compliance to treatment difficult
* Able to give informed consent

Exclusion Criteria:

* T3a or above
* Gleason 4+3=7
* PSA>20ng/ml

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must have prostate cancer
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with acute Radiation Oncology/ Toxicity Grading (RTOG) urinary toxicity | At 12 weeks post completion of treatment
  Clinician reported cumulative Grade 2 or worse RTOG acute GU toxicity from baseline up to 12 weeks post treatment (scale 0-4 with 0 being none increasing severity to grade 4).
The number of patients with acute Common Terminology for Adverse Events (CTCAE) urinary toxicity | At 12 weeks post completion of treatment
  Clinician reported cumulative Grade 2 or worse CTCAE v5.0 acute GU toxicity from baseline up to 12 weeks post treatment (scale 0-5 with increasing severity to death at grade 5)
The number of patients with acute Radiation Oncology/ Toxicity Grading (RTOG) bowel toxicity | At 12 weeks post treatment
  Clinician reported cumulative Grade 2 or worse RTOG acute GI toxicity from baseline up to 12 weeks post treatment (scale 0-4 with 0 being none increasing severity to grade 4).
The number of patients with acute Common Terminology for Adverse Events (CTCAE) bowel toxicity | At 12 weeks
  Clinician reported cumulative Grade 2 or worse CTCAE v5.0 acute GI toxicity from baseline up to 12 weeks post treatment (scale 0-5 with increasing severity to death at grade 5).

SECONDARY OUTCOMES:
The number of patients with late Radiation Oncology/ Toxicity Grading (RTOG) urinary toxicity | At 24 months post completion of radiotherapy treatment
  Clinician reported Grade 2 or worse RTOG late GU toxicity at 24 months (scale 0-4 with 0 being none increasing severity to grade 4).
The number of patients with late Common Terminology for Adverse Events (CTCAE) urinary toxicity | At 24 months post completion of radiotherapy treatment
  Clinician reported Grade 2 or worse CTCAE v5.0 late GU toxicity at 24 months (scale 0-5 with increasing severity to death at grade 5).
The number of patients with late Radiation Oncology/ Toxicity Grading (RTOG) bowel toxicity | At 24 months post completion of radiotherapy treatment
  Clinician reported Grade 2 or worse RTOG late GI toxicity at 24 months (scale 0-4 with 0 being none increasing severity to grade 4).
The number of patients with late Common Terminology for Adverse Events (CTCAE) bowel toxicity | At 24 months post completion of radiotherapy treatment
  Clinician reported Grade 2 or worse CTCAE v5.0 late GI toxicity at 24 months (scale 0-5 with increasing severity to death at grade 5).
Cumulative number of patients who experienced late Radiation Oncology/ Toxicity Grading (RTOG) urinary toxicity | From 6-24 months
  Clinician reported cumulative Grade 2 or worse RTOG late GU toxicity from 6 months to 24 months post treatment (scale 0-4 with 0 being none increasing severity to grade 4).
Cumulative number of patients who experience late Common Terminology for Adverse Events (CTCAE) urinary toxicity | From 6-24 months
  Clinician reported cumulative Grade 2 or worse CTCAE v5.0 late GU toxicity from 6 months to 24 months post treatment (scale 0-5 with increasing severity to death at grade 5).
Cumulative number of patients who experience late Radiation Oncology/ Toxicity Grading (RTOG) bowel toxicity | From 6-24 months
  Clinician reported cumulative Grade 2 or worse RTOG late GI toxicity from 6 months to 24 months post treatment (scale 0-4 with 0 being none increasing severity to grade 4).
Cumulative number of patients who experience late Common Terminology for Adverse Events (CTCAE) bowel toxicity | From 6-24 months
  Clinician reported cumulative Grade 2 or worse CTCAEv5.0 late GI toxicity from 6 months to 24 months post treatment (scale 0-5 with increasing severity to death at grade 5).
Quality of life patient reported outcome measure Expanded Prostate Index Composite-26 (EPIC-26) | Pre treatment to 24 months post treatment
  Expanded Prostate Index Composite-26 (EPIC-26), patient reported outcome measure of urinary, bowel, sexual, physical and mental health
Quality of life patient reported outcome measure International Prostate Symptom Score (IPSS) | Pre treatment to 24 months post treatment
  International Prostate Symptom Score (IPSS), a patient reported outcome measure of urinary bother
Quality of life patient reported outcome measure International Index of Erectile Function-5 (IIEF-5) | Pre treatment to 24 months post treatment
  International Index of Erectile Function-5 (IIEF-5), a patient reported outcome measure of erectile and sexual function
Quality of life patient reported outcome measure Vaizy Score | Pre treatment to 24 months post treatment
  Vaizey score, a patient reported assessment of bowel function

OTHER OUTCOMES:
Urethral dose sparing and acute Radiation Oncology/ Toxicity Grading (RTOG) | To be assessed at week 12 and month 24 post completion of treatment
  HypoCath Image Guidance with RayPilot and urethral dose sparing will result in lower grade 2+ RTOG GU acute toxicity than reported in the PACE-B trial when using a standard Linear accelerator
Urethral dose sparing and acute Common Terminology for Adverse Events (CTCAE) | To be assessed at week 12 and month 24 post completion of treatment
  HypoCath Image Guidance with RayPilot and urethral dose sparing will result in lower grade 2+ CTCAE v5.0 GU acute toxicity than reported in the PACE-B trial when using a standard Linear accelerator
Urethral dose sparing late Radiation Oncology/ Toxicity Grading (RTOG) | To be assessed at week 12 and month 24 post completion of treatment
  HypoCath Image Guidance with RayPilot and urethral dose sparing will result in lower grade 2+ RTOG GU late toxicity than reported in the PACE-B trial when using a standard Linear accelerator
Urethral dose sparing late Common Terminology for Adverse Events ( CTCAE | To be assessed at week 12 and month 24 post completion of treatment
  HypoCath Image Guidance with RayPilot and urethral dose sparing will result in lower grade 2+ CTCAE v5.0 GU late toxicity than reported in the PACE-B trial when using a standard Linear accelerator

CONTACTS AND LOCATIONS:
Overall Officials: Duncan B McLaren, MBBS, Principal Investigator — NHS Lothian & University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data generated is specific to using the RayPilot HypoCath System when delivering the treatment. Results will be presented and published but individual patient data would not be supplied